CLINICAL TRIAL: NCT03397394
Title: A Phase 2, Open-label Study of Rucaparib in Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: Rucaparib in Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Acronym: ATLAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efficacy did not meet the continuance criteria and DMC recommended to stop enrollment.
Sponsor: pharmaand GmbH (Industry)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-085; 2017-004166-10 (EudraCT Number)
Record Dates: First submitted 2017-12-21; First posted 2018-01-12 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Renal Pelvis Carcinoma; Ureter Carcinoma; Urinary Bladder Carcinoma; Urethra Carcinoma; Muscle Invasive Bladder Cancer
Keywords: PARP inhibitor; PARPi; HRD; ATLAS; homologous recombination; DNA repair; LOH; DNA defect; DNA anomaly; Rucaparib; MIBC
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Ureteral Neoplasms; Urethral Neoplasms | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rucaparib (Experimental): Oral rucaparib (monotherapy)
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — Rucaparib will be administered daily.
  Other Names: CO-338

SUMMARY:
The purpose of the ATLAS study is to determine how patients with locally advanced unresectable or metastatic urothelial carcinoma respond to treatment with rucaparib.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed locally advanced unresectable or metastatic transitional cell carcinoma of the urothelium (renal pelvis, ureter, urinary bladder or urethra)
* Received 1 or 2 prior treatment regimens for advanced or metastatic disease
* Confirmed radiologic disease progression during or following recent treatment
* Mandatory biopsy is required during screening
* Measurable disease per RECIST v1.1
* Adequate organ function
* ECOG 0 or 1

Exclusion Criteria:

* Prior treatment with a PARP inhibitor
* Symptomatic and/or untreated CNS metastases
* Duodenal stent and/or any gastrointestinal disorder that may interfere with absorption of rucaparib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (41):
  - Pinnacle Oncology, Honor Health, Scottsdale, Arizona
  - University of California San Diego (UCSD), Moores Cancer Center, La Jolla, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Universityof California, Irvine, Orange, California
  - Saint John's Health Center - John Wayne Cancer Institute (JWCI), Santa Monica, California
  - Stanford University School of Medicine, Stanford, California
  - Hartford Health Care Cancer Institute, Hartford, Connecticut
  - Eastern Connecticut Hematology & Oncology Associates (ECHO), Norwich, Connecticut
  - Medstar Georgetown University Medical Center, Washington D.C., District of Columbia
  - Miami Cancer Institute, Baptist Health South Florida, Miami, Florida
  - Northwestern University, Chicago, Chicago, Illinois
  - Indiana University - Melvin and Bren Simon Cancer Center (IUSCC), Indianapolis, Indiana
  - The University of Iowa and Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Cancer Center, Louisville, Kentucky
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - University of Maryland, Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota Oncology Hematology P.A. (USO - US Oncology), Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada (CCCN), Las Vegas, Nevada
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico UNM Cancer Research and Treatment Center, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C. (USO - US Oncology), Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York - Presbyterian Hospital-Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Duke Cancer Institute, Durham, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Northwest Cancer Specialists P.C. (USO - US Oncology), Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Atlantic Urology Clinics, Myrtle Beach, South Carolina
  - University Oncology & Hematology, Chattanooga, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Texas Oncology PA (USO - US Oncology), Dallas, Texas
  - University of Texas, UT Health Science Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Emily Couric Clinical Center, Charlottesville, Virginia
  - University of Washington / Seattle Cancer Care Alliance, Seattle, Washington
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin
- France (5):
  - Centre de Lutte Contre le Cancer (CLCC) - Universite de Lyon - Centre Leon-Berard, Lyon
  - Hopital Saint-Louis, Paris
  - Centre de Lutte Contre le Cancer - Institut de Cancerologie de l'Ouest - Rene Gauducheau, Saint-Herblain
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Urologische und Kinderurologische Universitätsklinik im Malteser, Erlangen
  - Universitatsklinikum Munster / Urologie und Kinderurologie, Münster
  - Studienpraxis Urologie, Nürtingen
- Italy (4):
  - Fondazionerca sul Cancro ONLUS - Istituto di Candiolo IRCCS, Candiolo
  - IRCCS Ospedale San Raffaele - Medical Oncology Dept, Milan
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Azienda Ospedaliera Universitaria Federico II Oncologia Medica, Naples
- Spain (9):
  - Universidad de Navarra - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Clinica Universitaria de Navarra Madrid, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
- United Kingdom (2):
  - Sarah Cannon Research Institute - United Kingdom - London Office, London
  - Guy's & St. Thomas' Hospital (London Oncology Clinic), London

REFERENCES:
- [Derived] Grivas P, Loriot Y, Morales-Barrera R, Teo MY, Zakharia Y, Feyerabend S, Vogelzang NJ, Grande E, Adra N, Alva A, Necchi A, Rodriguez-Vida A, Gupta S, Josephs DH, Srinivas S, Wride K, Thomas D, Simmons A, Loehr A, Dusek RL, Nepert D, Chowdhury S. Efficacy and safety of rucaparib in previously treated, locally advanced or metastatic urothelial carcinoma from a phase 2, open-label trial (ATLAS). BMC Cancer. 2021 May 24;21(1):593. doi: 10.1186/s12885-021-08085-z. PMID 34030643

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 97 subjects were recruited from 40 sites across 6 countries.
Groups:
- HRD Unknown: Patients with HRD status unknown who received continuous dosing with rucaparib 600 mg twice a day (BID) in 28-day cycles. Patients whose tumor genome-wide LOH was not tested or not determined were considered HRD unknown.
- HRD Negative: Patients with HRD status negative who received continuous dosing with rucaparib 600 mg twice a day (BID) in 28-day cycles. Patients whose tumor had genome-wide LOH < 10% were considered HRD-negative.
- HRD Positive: Patients with HRD status positive who received continuous dosing with rucaparib 600 mg twice a day (BID) in 28-day cycles. Patients whose tumor had genome-wide LOH ≥ 10% were considered HRD-positive.
Period: Overall Study
Arm/Group | HRD Unknown | HRD Negative | HRD Positive
Started | 47 | 30 | 20
Completed | 47 | 30 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HRD Unknown | HRD Negative | HRD Positive | Total
Number analyzed (Participants) | 47 | 30 | 20 | 97
Age, Continuous [Median (Full Range); unit: years] | 66.0 [50 to 85] | 66.0 [47 to 85] | 71.0 [39 to 87] | 66.0 [39 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 9 | 21
  Male | 38 | 27 | 11 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 1 | 12
  Not Hispanic or Latino | 29 | 23 | 17 | 69
  Unknown or Not Reported | 11 | 3 | 2 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 2 | 0 | 3
  White | 32 | 24 | 18 | 74
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 3 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per RECIST Version 1.1
Description: ORR is defined as the proportion of patients with a confirmed response of complete response (CR) or partial response (PR) by RECIST v1.1 as assessed by the investigator. Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR), is at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: Time from first dose to date of progression, up to approximately 19 months
Population: Intent-to-treat Population (ITT) with measurable disease at Baseline - The ITT population includes all patients who received at least 1 dose of rucaparib. One patient each in the HRD negative and HRD positive groups did not have measurable disease at Baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: All patients
Arm/Group | HRD Unknown | HRD Negative | HRD Positive | Overall
Number analyzed (Participants) | 47 | 29 | 19 | 95
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Progression-free Survival (PFS) According to RECIST v1.1, as Assessed by the Investigator
Description: PFS is calculated as 1+ the number of days from the first dose of study drug to disease progression by RECIST, as determined by the investigator or death due to any cause, whichever occurs first.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 10 months
Population: Intent-to-Treat population - all patients who received at least 1 dose of rucaparib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HRD Unknown | HRD Negative | HRD Positive | Overall
Number analyzed (Participants) | 47 | 30 | 20 | 97
months | 1.8 [1.6 to 2.0] | 1.8 [1.5 to 2.0] | 1.4 [1.2 to 3.6] | 1.8 [1.6 to 1.9]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as time from the date of first dose of rucaparib to the date of death due to any cause. Patients without a known date of death were to be censored on the date the patient was last known to be alive. A Kaplan-Meier analysis of OS was planned, however, due to early study termination and limited duration of OS follow-up, a descriptive summary of total deaths are presented. This includes deaths recorded on study (from first dose of study drug until 28 days after last dose of study drug), and deaths recorded in long-term follow-up (from last dose +28 days until death, loss to follow-up, withdrawal of consent, or study closure).
Time Frame: The total study time for reporting of deaths was approximately 19 months.
Population: Intent-to-Treat population - all patients who received at least 1 dose of rucaparib
Measure: Count of Participants; unit: Participants
Arm/Group | HRD Unknown | HRD Negative | HRD Positive | Overall
Number analyzed (Participants) | 47 | 30 | 20 | 97
Participants | 15 | 15 | 9 | 39

4. Secondary Outcome: Pharmacokinetics - Trough (Cmin) Level Rucaparib Concentrations
Description: Plasma were collected for trough level PK analysis of rucaparib 1 hour before the morning dose on Cycle 2 Day 1, Cycle 3 Day 1, and Cycle 4 Day 1.
Time Frame: From Cycle 2 Day 1 to Cycle 4 Day 1, or approximately 2 months
Population: Safety population - all patients who received at least 1 dose of rucaparib and who had at least 1 PK sample collected. The number analyzed at each timepoint includes only those participants who remained on study and with viable samples collected at that timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HRD Unknown | HRD Negative | HRD Positive | Overall
Number analyzed (Participants) | 24 | 13 | 10 | 47
ng/mL
  Cycle 2 Day 1 | 2354.03 (2173.055) | 1927.77 (1352.707) | 1853.84 (1533.622) | 2129.70 (1831.099)
  Cycle 3 Day 1: number analyzed (Participants) | 10 | 6 | 2 | 18
  Cycle 3 Day 1 | 2037.90 (1253.715) | 1331.17 (357.010) | 643.00 (688.722) | 1647.33 (1068.270)
  Cycle 4 Day 1: number analyzed (Participants) | 4 | 5 | 2 | 11
  Cycle 4 Day 1 | 2225.00 (763.348) | 2058.00 (705.280) | 1585.00 (487.904) | 2032.73 (672.891)

ADVERSE EVENTS:
Time Frame: Adverse events for each patient were reported from the first dose until 28 days after last dose of study drug, and the total study time for adverse event reporting was approximately 19 months.
Arm/Group | HRD Unknown | HRD Negative | HRD Positive | Overall
All-Cause Mortality (participants affected / at risk) | 9/47 | 8/30 | 7/20 | 24/97
Serious Adverse Events (participants affected / at risk) | 20/47 | 14/30 | 11/20 | 45/97
Other Adverse Events (participants affected / at risk) | 45/47 | 29/30 | 19/20 | 93/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HRD Unknown (N=47) | HRD Negative (N=30) | HRD Positive (N=20) | Overall (N=97)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 5
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 2
Pyelonephritis (Infections and infestations) | 2 | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 9 | 3 | 18
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HRD Unknown (N=47) | HRD Negative (N=30) | HRD Positive (N=20) | Overall (N=97)
Anaemia (Blood and lymphatic system disorders) | 16 | 10 | 8 | 34
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 6 | 3 | 14
Abdominal pain (Gastrointestinal disorders) | 4 | 5 | 2 | 11
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 3 | 4
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 10 | 5 | 5 | 20
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 1 | 12
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 0 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 26 | 9 | 6 | 41
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 2 | 3
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 13 | 6 | 3 | 22
Asthenia (General disorders) | 12 | 4 | 1 | 17
Chest pain (General disorders) | 1 | 2 | 0 | 3
Chills (General disorders) | 1 | 0 | 1 | 2
Fatigue (General disorders) | 21 | 12 | 7 | 40
Localized oedema (General disorders) | 0 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 1 | 1 | 2 | 4
Nodule (General disorders) | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 3 | 1 | 4 | 8
Pain (General disorders) | 4 | 3 | 1 | 7
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 4 | 2 | 3 | 9
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 1 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1 | 2
Sialoadenitis (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 4 | 3 | 3 | 10
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 4
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 6 | 2 | 3 | 11
Aspartate aminotransferase increased (Investigations) | 5 | 5 | 5 | 15
Blood alkaline phosphatase increased (Investigations) | 3 | 2 | 0 | 5
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 6 | 11 | 4 | 21
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 2 | 3
Neutrophil count decreased (Investigations) | 1 | 0 | 2 | 3
Platelet count decreased (Investigations) | 2 | 3 | 3 | 8
Transaminases increased (Investigations) | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 6 | 7 | 0 | 13
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 14 | 7 | 7 | 28
Dehydration (Metabolism and nutrition disorders) | 5 | 4 | 1 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 3 | 1 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 5 | 0 | 1 | 6
Dysgeusia (Nervous system disorders) | 8 | 7 | 1 | 16
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | 2
Somnolence (Nervous system disorders) | 3 | 0 | 1 | 4
Insomnia (Psychiatric disorders) | 7 | 2 | 1 | 10
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 1 | 3
Haematuria (Renal and urinary disorders) | 1 | 4 | 1 | 6
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 1 | 12
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 3
Hypertension (Vascular disorders) | 3 | 0 | 0 | 3
Intermittent claudication (Vascular disorders) | 0 | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2

LIMITATIONS AND CAVEATS:
The study was terminated early based on an interim analysis by the Data Monitoring Committee that demonstrated that ORR did not meet the protocol-defined continuance criteria. There were no confirmed responses observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT03397394/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT03397394/SAP_001.pdf